CLINICAL TRIAL: NCT06029816
Title: A Single-arm, Open-label, Multicenter Phase II Clinical Study of Neratinib Tablets in the Treatment of Advanced NSCLC With Rare EGFR Mutations
Brief Title: Neratinib Tablets in the Treatment of Advanced NSCLC With Rare EGFR Mutations
Acronym: CVL009-2001
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Convalife (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVL009-2001; Chinadrugtrials (Other: CTR20231827)
Record Dates: First submitted 2023-07-31; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: NSCLC
Keywords: NSCLC; EGFR; Neratinib tablets
MeSH Terms: interventions — neratinib

STUDY DESIGN:
Intervention Model Description: Fourteen patients each had three mutation sites and 42 patients were co-enrolled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm1-Exon 18 (Experimental): Exon 18 G719X, E709X, etc，Up to 14 patients will be enrolled in this group and will be treated with neratinib tablets in 28-day cycles，
  Interventions: Drug: Neratinib tablets
- Arm2-Exon 20 (Experimental): S768I in exon 20，Up to 14 patients will be enrolled in this group and will be treated with neratinib tablets in 28-day cycles，
  Interventions: Drug: Neratinib tablets
- Arm3-Exon 21 (Experimental): L861Q of exon 21，Up to 14 patients will be enrolled in this group and will be treated with neratinib tablets in 28-day cycles，
  Interventions: Drug: Neratinib tablets

INTERVENTIONS:
Drug: Neratinib tablets — Neratinib tablets
  Other Names: Epilepsy

SUMMARY:
Single-arm, open-label, multicenter phase II clinical study

DETAILED DESCRIPTION:
Fourteen patients each had three mutation sites and 42 patients were co-enrolled，To evaluate the objective response rate (ORR) of neratinib Tablets in advanced NSCLC with rare EGFR mutations (including G719X, E709X in exon 18, S768I in exon 20 and L861Q in exon 21).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Histologically or cytologically confirmed non-small cell lung cancer, stage IIIB or IV according to IASLC 2009;
3. Tissue or blood samples are confirmed by the central laboratory or research center as rare EGFR mutations, including exon 18 G719X, E709X, etc., S768I in exon 20 and at least one of the L861Q mutations in exon 21;
4. Ineffective or intolerant to standard treatment regimens, and disease progression after treatment;
5. The number of previous chemotherapy regimens does not exceed 2 (a. replacement of platinum drugs for drug toxicity reasons is counted as a regimen; b. postoperative adjuvant chemotherapy, from the end of treatment to recurrence > 6 months is not counted as a previous chemotherapy regimen);
6. ECOG standard score 0-1;
7. Predicted survival ≥ 12 weeks;
8. Presence of measurable lesions according to RECIST 1.1: At least one lesion that is not irradiated, ≥ 10 mm in long diameter (lymph node lesions need to be ≥ 15 mm in short diameter), and can be accurately measured at baseline and can be repeatedly measured under CT or MRI; If the subject only has post-radiotherapy lesion, and this lesion has been confirmed as imaging progression and can be measured, it can be selected as target lesion (except for brain lesion), and brain lesion is not included as measurable target lesion;
9. Subjects with asymptomatic brain metastases or brain metastases can be included in this study when the following conditions are met: brain metastases are treated and stable, such as clinical examination and brain scan (MRI or CT scan) confirmed at least 4 no evidence of lesion progression during the screening period, no neurological symptoms and no need for corticosteroid therapy. If the subject has brain metastases that have been treated surgically or with radiation, a time window of ≥ 4 weeks is required before the first dose of nelatidine tablets to ensure that adverse events associated with radiation or surgical treatment have decreased to ≤ Grade 1;
10. Bone marrow reserve or organ function needs to meet the following laboratory value criteria:

    * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L
    * Platelet count (PLT) ≥ 90 × 109/L
    * Hemoglobin (Hb) ≥ 90 g/L
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN; ≤ 5 × ULN in the presence of liver metastases
    * Serum total bilirubin (TBIL) ≤ 1.5 × ULN
    * Blood urea nitrogen/urea nitrogen (UREA/BUN) and creatinine (Cr) ≤ 1.5 × ULN
    * Coagulation international normalized ratio (INR) ≤ 1.5 ULN and APTT ≤ 1.5 ULN;
    * Urine protein < 2 + (when baseline urine protein is 2 +, 24-hour urine protein quantification should be performed, and inclusion can only be made when ≤ 1 g) * ULN = upper limit of normal
11. Women of childbearing potential should agree to take contraceptive measures (such as intrauterine device, contraceptive or condom) during the study and within 6 months after the end of the study; 7. Blood pregnancy test is negative before enrollment and patients must be non-lactating; men should agree to take contraceptive measures during the study and within 6 months after the end of the study;
12. Patients voluntarily participate in this study, sign the informed consent form, and have good compliance.

Exclusion Criteria:

1. Received any of the following treatments: 1. previous treatment with any EGFR tyrosine kinase inhibitor; 2. major surgery 4 times before the first dose of the study drug; c. 4 times before the first dose of the study drug, more than 30% of bone marrow irradiation, or extensive radiotherapy; d. within 7 days before the first dose of the study drug, the use of CYP3A4 strong inhibitors, inducers or drugs that are CYP3A4 sensitive substrates with a narrow therapeutic window;
2. Patients with other malignant tumors and need standard treatment or major surgery within 2 years after the first dose of study treatment;
3. In the beginning of the study treatment, there are greater than CTCAE grade 1 failed to alleviate the residual toxicity of previous treatment, except alopecia and previous chemotherapy-induced grade 2 neurotoxicity;
4. Spinal cord compression or brain metastasis, unless asymptomatic, stable condition, and not requiring steroid therapy for at least 2 weeks before the first dose of study treatment;
5. Poor blood pressure control after drug treatment (systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 100 mmHg);
6. Patients with severe or uncontrollable systemic diseases, including gastrointestinal ulcers and bleeding and other diseases;
7. There are many factors that affect the oral administration of drugs (such as inability to swallow, chronic diarrhea, intestinal obstruction and other gastrointestinal diseases or abnormalities);
8. 12 ECG: QTcF: female > 470 ms, male > 450 ms;
9. Echocardiography: score (LVEF) ≤ 50%;
10. History of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid therapy or any evidence of clinically active interstitial lung disease;
11. History of immunodeficiency, including HIV test positive, active hepatitis B/C (HBV-DNA > 1000 IU/mL or > 2500 copies/mL, HCV-RNA ≥ 10 ³ copies/mL) or suffering from other acquired, congenital immunodeficiency diseases, or history of organ transplantation;
12. Women who are lactating or have a positive pregnancy test result before the first dose of study treatment;
13. 4 Participated in any other drug clinical study before the first dose;
14. The investigator judges that there are any patients who endanger the patient's safety, interfere with the study assessment, and have poor compliance;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-11-20 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
IRC-assessed objective response rate (ORR) | Through study completion, an average of 1 year
  IRC-assessed objective response rate (ORR)

OTHER OUTCOMES:
ORR by investigator | Through study completion, an average of 1 year
  ORR by investigator
Overall Survival (OS) | Through study completion, an average of 1 year
  Overall Survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Wenfeng Fang, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No